CLINICAL TRIAL: NCT06209697
Title: Isoflavones Obtained From Red Clover Improves Both Dyslipidemia and Menopausal Symptoms in Menopausal Women: a Prospective Randomized Placebo-controlled Trial
Brief Title: Effect of Red Clover on Menopause Symptoms and Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ece Yigit, Principal Investigator / Asst. Prof. Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: redclover*
Record Dates: First submitted 2023-12-14; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Menopause
Keywords: menopause, hyperlipidemia, red clover
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: The study included postmenopausal women who had naturally entered menopause and had applied to the outpatient clinics of Istanbul Medipol University Internal Medicine or Gynecology Departments with symptoms of menopause. Other inclusion criteria were: having a history of amenorrhea for at least 12 months, being aged 45-55, having received a diagnosis of dyslipidemia (at the present admission or within the past 3 months), not receiving treatment for dyslipidemia, absence of other chronic diseases, having a follicle stimulating hormone level of >40 pg/mL and having a body mass index (BMI) of <30 kg/m2.The subjects were divided into two groups: red clover and placebo groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For the randomization process, patients were provided with slips of paper bearing numbers starting from 1, assigned based on the order of admission by the admitting physician. Subsequently, they were directed to the appropriate nurse. The outpatient clinic nurse assigned red clover treatment to subjects with an odd-numbered slip and placebo to those with an even-numbered slip. The nurse documented the medication assigned to each patient, while the researchers and subjects remained blinded to this information
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- red clover (Active Comparator): Red clover (Promensil, PharmaCare Europe Ltd., UK) and placebo (starch capsules) were administered orally twice a day with an interval of 12 hours for a total period of 6 months. Red clover capsules contained 40 mg of standardized red clover isoflavones in each capsule [genistein (1 mg), daidzein (1 mg), biochanin A (23 mg) and biochanin B (formononetin, 15 mg)].
  Interventions: Dietary Supplement: red clover
- placebo (Placebo Comparator): Placebo capsules were ordered to be prepared with the same color, taste and smell as the red cover capsules. Placebo capsules were administered orally twice a day with an interval of 12 hours for a total period of 6 months.
  Interventions: Dietary Supplement: red clover

INTERVENTIONS:
Dietary Supplement: red clover — Red clover (Promensil, PharmaCare Europe Ltd., UK) and placebo (starch capsules) were administered orally twice a day with an interval of 12 hours for a total period of 6 months.

SUMMARY:
The goal of this clinical trial is to investigate the effects of red clover isoflavones on menopausal symptoms and lipid profile in menopausal females.This prospective randomized, double-blind, placebo-controlled study included postmenopausal women with dyslipidemia. The red clover group received 40 mg isoflavone red clover capsule twice daily for 6 months, while placebo was 40 mg starch capsules, twice daily. Data were collected at baseline, 3 months and 6 months. The study was completed with 75 subjects [red clover (n = 39), placebo (n = 36)]. Menopause Rating Scale (MRS) was applied to calculate subdimension and total scores. Blood lipid profile, including total cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglyceride levels were measured.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the effects of red clover isoflavones on menopausal symptoms and lipid profile in menopausal females. This was a prospective, randomized, double-blind, placebo-controlled study conducted between March 2022 and September 2023 in the Departments of Gynecology and Internal Medicine of Medipol University Hospital, Istanbul, Turkey. The subjects were divided into two groups: red clover and placebo groups. For the randomization process, patients were provided with slips of paper bearing numbers starting from 1, assigned based on the order of admission by the admitting physician. Subsequently, they were directed to the appropriate nurse. The outpatient clinic nurse assigned red clover treatment to subjects with an odd-numbered slip and placebo to those with an even-numbered slip. The nurse documented the medication assigned to each patient, while the researchers and subjects remained blinded to this information. Red clover (Promensil, PharmaCare Europe Ltd., UK) and placebo (starch capsules) were administered orally twice a day with an interval of 12 hours for a total period of 6 months. Red clover capsules contained 40 mg of standardized red clover isoflavones in each capsule [genistein (1 mg), daidzein (1 mg), biochanin A (23 mg) and biochanin B (formononetin, 15 mg)]. Placebo capsules were ordered to be prepared with the same color, taste and smell as the red cover capsules. The patients' total cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglyceride levels were measured using the enzymatic colorimetric method (Hitachi 747 autoanalyzer; Germany) from antecubital venous blood samples taken at 8 AM after a 12-hour overnight fast at baseline, at 3-month follow-up and at 6-month follow-up. The severity of menopausal symptoms was assessed utilizing the Menopause Rating Scale (MRS). Data were collected at baseline, 3 months and 6 months. The study was completed with 75 subjects [red clover (n = 39), placebo (n = 36)].

ELIGIBILITY:
Inclusion Criteria:

History of amenorrhea for at least 12 months

Being aged 45-55

Having received a diagnosis of dyslipidemia (at the present admission or within the past 3 months)

Not receiving treatment for dyslipidemia

Absence of other chronic diseases

Follicle stimulating hormone level of >40 pg/mL

Body mass index (BMI) of <30 kg/m2

Exclusion Criteria:

Currently or previously undergoing hormone replacement therapy (either in the past, immediately before, or during the study)

Using any phytotherapeutic drug

Diagnosed with diabetes

Presence of anemia

Presence of cardiovascular disease Presence of musculoskeletal disease

Presence of asthma / chronic obstructive pulmonary disease

Presence of malignancy

Prsence of genital or gynecological disease (excluding menopausal symptoms)

Presence of neurological or psychiatric disease

Conditions involving acute or chronic inflammation

Experiencing acute or chronic infection

Displaying abnormal liver, kidney, or thyroid function tests

Engaging in smoking, alcohol consumption, or drug use

Suffering from sexual dysfunction (except for menopause-related reasons)

Unable to complete the study, or not attending 3-month or 6-month follow-up

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study evaluates women in the postmenopausal period.
Enrollment: 82 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures were to assess the differences in MRS scores (somatic, psychological, urogenital and total score) and lipid profile (total cholesterol, LDL-C, HDL-C and triglyceride levels). | 6 months
  The patients' total cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglyceride levels were measured using the enzymatic colorimetric method (Hitachi 747 autoanalyzer; Germany) from antecubital venous blood samples taken at 8 AM after a 12-hour overnight fast at baseline, at 3-month follow-up and at 6-month follow-up. Values of the lipid profile were measured in mg/dl. The severity of menopausal symptoms was assessed utilizing the Menopause Rating Scale (MRS). MRS is a questionnaire consisting of 11 questions under 3 main categories, namely, the somatic disorders, psychological disorders, urogenital disorders. Each question is scored as 0 (no complaints), 1 (mild), 2 (moderate), 3 (severe) and 4 (very severe) based on the perceived severity of respondents.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Pendik /Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
MRS results and laboratory data can be shared while protecting patients' personal data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Shakeri F, Taavoni S, Goushegir A, Haghani H. Effectiveness of red clover in alleviating menopausal symptoms: a 12-week randomized, controlled trial. Climacteric. 2015;18(4):568-73. doi: 10.3109/13697137.2014.999660. Epub 2015 Feb 24. PMID 25581426
- [Result] Kanadys W, Baranska A, Blaszczuk A, Polz-Dacewicz M, Drop B, Kanecki K, Malm M. Evaluation of Clinical Meaningfulness of Red Clover (Trifolium pratense L.) Extract to Relieve Hot Flushes and Menopausal Symptoms in Peri- and Post-Menopausal Women: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2021 Apr 11;13(4):1258. doi: 10.3390/nu13041258. PMID 33920485
- [Result] Luis A, Domingues F, Pereira L. Effects of red clover on perimenopausal and postmenopausal women's blood lipid profile: A meta-analysis. Climacteric. 2018 Oct;21(5):446-453. doi: 10.1080/13697137.2018.1501673. PMID 30269660
- [Result] Hidalgo LA, Chedraui PA, Morocho N, Ross S, San Miguel G. The effect of red clover isoflavones on menopausal symptoms, lipids and vaginal cytology in menopausal women: a randomized, double-blind, placebo-controlled study. Gynecol Endocrinol. 2005 Nov;21(5):257-64. doi: 10.1080/09513590500361192. PMID 16373244
- [Result] Campbell MJ, Woodside JV, Honour JW, Morton MS, Leathem AJ. Effect of red clover-derived isoflavone supplementation on insulin-like growth factor, lipid and antioxidant status in healthy female volunteers: a pilot study. Eur J Clin Nutr. 2004 Jan;58(1):173-9. doi: 10.1038/sj.ejcn.1601764. PMID 14679383